CLINICAL TRIAL: NCT05242367
Title: A Randomized, Double Blind Sham Controlled Clinical Trial to Evaluate the Efficacy of Electrical Vestibular Nerve Stimulation (VeNS), Compared to a Sham Control for Treatment of Post- Traumatic Stress Disorder (PTSD)
Brief Title: Electrical Vestibular Nerve Stimulation (VeNS) as a Treatment for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: University of California, San Diego (Other); Clinical Trial Mentors (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS003
Record Dates: First submitted 2022-02-09; First posted 2022-02-16 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active VeNS (Active Comparator): The active device utilizes a technology termed vestibular nerve stimulation (VeNS). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Interventions: Device: Modius Spero active device
- Sham VeNS (Sham Comparator): The sham device looks identical to the active device and interacts with the app in a similar manner to the active device. It will apply some stimulation to a user for a limited period of time (30 seconds), before tapering down to zero over a further 20 seconds, thus creating the impression of an active device. The device will be placed on the head in a manner analogous to headphones with hydrogel electrodes placed over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Modius Spero active device — Battery powered non-invasive neurostimulation device
  Arms: Active VeNS
Device: Sham device — Placebo comparator sham device (no active stimulation)
  Arms: Sham VeNS

SUMMARY:
Trial title: A Randomized, Double Blind Sham Controlled Clinical Trial to Evaluate the Efficacy of Electrical Vestibular Nerve Stimulation (VeNS), Compared to a Sham Control for Treatment of PTSD

The aim of this study: To better evaluate the efficacy of non-invasive electrical vestibular nerve stimulation (VeNS) as a method of treating PTSD, as compared to a sham control.

Allocation: Randomized to either active device or control device usage.

Endpoint classification: Efficacy Study Intervention Model: Parallel Assignment in 1:1 active to control allocation

Sample size: The aim is to recruit a total of up to 400 participants. The study will last 12 weeks in total for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosed PTSD by a medical practitioner
* Post-Traumatic Checklist (PCL-5) score or 31 or above
* Eligibility confirmed via the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
* Male or female, age ≥ 22 years and ≤ 80 years at the time of signing informed consent
* Ability and willingness to complete all study visits and procedures, including completion of mental health questionnaires
* Ability and willingness to adhere to 30 minutes usage of the device daily for the duration of the trial
* Agreement not to start any new PTSD, mental health, or insomnia medications for the duration of the trial and/or to inform the study team if intending on starting any new PTSD, mental health, or insomnia medications
* Agreement not to change any PTSD specific treatments for the duration of the trial e.g cognitive processing therapy
* Agreement not to undergo any significant lifestyle changes that may affect sleep (e.g. excessive exercise, sleep interventions etc.) for the duration of the trial
* Agreement not to use sleep trackers (e.g. Fitbit) for the duration of the trial
* Agreement not to travel across different time zones for the duration of the trial
* Access to Wi-Fi (for app to be able to upload usage data)
* Access to computer, laptop, iPad or tablet (to conduct remote study visits and complete study questionnaires remotely)
* Screening review by PTSD physician (study PI)
* Willingness to download and use a video platform (e.g Zoom) to conduct remote study visits
* Willingness to engage weekly with your Clinical Trial Mentor (CTM)

Exclusion Criteria:

* History of skin breakdown, eczema, or other dermatological condition (e.g., psoriasis) affecting the skin behind the ears
* History of severe tinnitus or vertigo
* History or presence of malignancy within the last year
* Use of beta-blockers within 1 month of starting the study
* History of chronic viral infection that causes vestibular neuropathy (e.g., hepatitis or HIV)
* Use of antihistamines
* A history of stroke or severe head injury as defined by a head injury that required a craniotomy or endotracheal intubation (in case this damaged the neurological pathways involved in vestibular stimulation)
* Taking H2-receptor antagonist medication
* Presence of permanently implanted battery powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator etc.)
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using an adequate contraceptive method
* Diagnosis of epilepsy
* Diagnosis of active migraines
* Previous use of Modius device
* Participation in other research studies sponsored by Neurovalens
* Participation in any other PTSD studies
* Not fluent in English language
* Have a member of the same household who is currently participating in this study
* Failure to agree to use of device daily during study participation
* Any other medical condition, or medication use, that in the opinion of the PI is likely to make the subject refractory to VeNS.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist PCL-5 score | 12 weeks
  To evaluate the effect of the Modius Sleep device, relative to control group, on the symptoms of PTSD, quantified by change in the PCL-5 Score.

SECONDARY OUTCOMES:
36-Item Short Form Survey (SF-36) score | 12 weeks
  To evaluate the effect of the Modius Spero device, relative to control group, on quality of life quantified by change in SF-36 score.
Generalised Anxiety Disorder (GAD-7) score | 12 weeks
  To evaluate the effect of the Modius Spero device, relative to control group, on anxiety, quantified by change in the GAD-7 score. GAD-7 is a self-report rating scale assessing the severity of anxiety (range 0-21), with higher score indicating more severe anxiety.
Insomnia Severity Index (ISI) score | 12 weeks
  To evaluate the effect of the Modius Spero device, relative to control group, on participants with insomnia. ISI is a self-report rating scale assessing the severity of insomnia symptoms (range 0-28) with higher scores indicating a more severe insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Colvonen, MD, Principal Investigator — UC San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided